CLINICAL TRIAL: NCT03615989
Title: Does Milk Augment the Acute Effect of Exercise on Bone Turnover and Inflammation
Brief Title: The Combined Effect of Dairy and Exercise on Bone and Inflammation
Acronym: Cre-Ex-Inf
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: York University (Other)
Collaborators: Brock University (Other)
Responsible Party: Principal Investigator, Andrea Josse, Assistant Professor, York University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-045; REB 17-402 (Other: Brock University)
Record Dates: First submitted 2018-07-30; First posted 2018-08-06 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Healthy; Females; Bone; Inflammation
Keywords: Bone Health; Females; Dairy; Exercise; Inflammation
MeSH Terms: conditions — Inflammation; Motor Activity | interventions — Plyometric Exercise; Carbohydrates; Water; Milk

STUDY DESIGN:
Intervention Model Description: Randomized acute Crossover Trial
Who Masked: Outcomes Assessor
Masking Description: Those completing the analyses were masked to the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise and Carbohydrate (CHO) (Placebo Comparator): Participants had a fasted, baseline blood sample (10ml) taken upon arrival to the lab. They then completed a supervised resistance and plyometric exercise bout. Immediately following exercise, 50g of carbohydrate (maltodextrin) + water was consumed. Two more blood samples followed the exercise bout at 5 minutes post (10ml) and 1 hour post (10ml). An additional 50g of carbohydrate was consumed with water 1 hour post exercise. Two more fasting blood samples (10ml) were taken 24 and 48 hours later.
  Interventions: Behavioral: Resistance and Plyometric Exercise; Dietary Supplement: Carbohydrate (Maltodextrin powder mixed with water)
- Exercise and Milk (Milk) (Experimental): Participants had a fasted, baseline blood sample (10ml) taken upon arrival to the lab. They then completed a supervised resistance and plyometric exercise bout. Immediately following exercise, ~500 ml of skim milk was consumed. Two more blood samples followed the exercise bout at 5 minutes post (10ml) and 1 hour post (10ml). An additional 500 ml of skim milk was consumed 1 hour post exercise. Two more fasting blood samples (10ml) were taken 24 and 48 hours later.
  Interventions: Behavioral: Resistance and Plyometric Exercise; Dietary Supplement: Skim Milk

INTERVENTIONS:
Behavioral: Resistance and Plyometric Exercise — A single resistance and plyometric exercise bout per trial.
Dietary Supplement: Carbohydrate (Maltodextrin powder mixed with water) — 50 grams immediately after exercise bout. 50 grams 1 hour after exercise bout.
  Other Names: CHO
  Arms: Exercise and Carbohydrate (CHO)
Dietary Supplement: Skim Milk — 500 ml immediately after exercise bout. 500 ml 1 hour after exercise bout.
  Other Names: Milk
  Arms: Exercise and Milk (Milk)

SUMMARY:
This study analyzes whether dairy supplementation positively impacts loading exercise-induced bone cell activity and inflammation in healthy young females.

DETAILED DESCRIPTION:
Introduction: Two million individuals at a cost of around 2.3 billion dollars a year in Canada suffer from osteoporosis. Research that emphasizes the treatment of this disease is important, but so is research that focuses on prevention; reducing bone loss and/or increasing bone mass when young. In addition, inflammation is an issue as it strongly relates to chronic disease. Countermeasures to improve bone health and inflammation, such as nutrition and exercise, should be explored and implemented. The proposed research combines both nutrition and exercise along with the assessment of bone turnover markers and inflammation in healthy young females, and aims to determine whether dairy versus a carbohydrate-based beverage positively impacts acute bone turnover and the inflammatory response following a bout of resistance and plyometric exercise.

Design: Randomized controlled crossover trial.

Participants: 13 healthy university aged females.

Methods: Participants were asked to complete 2 different acute exercise and nutritional supplement trials. Each trial will be assigned in random order. The two trials were: 1) exercise+carbohydrate (CHO), and 2) exercise+milk (Milk). The whole study, per participant, took a maximum of 8-12 weeks to complete as each supplement trial was separated by ~4 weeks. Each treatment is outlined below.

******DUE TO COVID-19, we removed the treatment trial which involved milk+creatine supplementation. Despite randomization, and before the trial was closed, only 11 participants completed this trial********

Anticipated Results: The investigators anticipate that dairy and exercise will have a greater positive impact on acute bone cell activity and inflammation in healthy young females compared to exercise and CHO.

ELIGIBILITY:
Inclusion Criteria:

* Female between the ages of 18 and 30 years
* Normal BMI (18.5-24.9) kg/m2
* Low to moderately physically active (0-2 times/week)
* No allergy to dairy protein or lactose intolerance
* On no medication related to a chronic condition
* On birth control (or not but with regular mensural cycle)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-14 (Actual)

PRIMARY OUTCOMES:
Acute Bone Cell Activity | Baseline
  Bone markers (OPG, RANKL, OC) measured in serum/plasma.
Acute Bone Cell Activity | Baseline
  Bone markers (SOST) measured in serum/plasma.
Acute Bone Cell Activity | Baseline
  Bone markers (CTX) measured in serum/plasma.
Acute Bone Cell Activity | 5 minutes post exercise
  Bone markers (OPG, RANKL, OC) measured in serum/plasma.
Acute Bone Cell Activity | 5 minutes post exercise
  Bone markers (SOST) measured in serum/plasma.
Acute Bone Cell Activity | 5 minutes post exercise
  Bone markers (CTX) measured in serum/plasma.
Acute Bone Cell Activity | 1 hour post exercise
  Bone markers (OPG, RANKL, OC) measured in serum/plasma.
Acute Bone Cell Activity | 1 hour post exercise
  Bone markers (SOST) measured in serum/plasma.
Acute Bone Cell Activity | 1 hour post exercise
  Bone markers (CTX) measured in serum/plasma.
Acute Bone Cell Activity | 24 hours post exercise
  Bone markers (OPG, RANKL, OC) measured in serum/plasma.
Acute Bone Cell Activity | 24 hours post exercise
  Bone markers (SOST) measured in serum/plasma.
Acute Bone Cell Activity | 24 hours post exercise
  Bone markers (CTX) measured in serum/plasma.
Acute Bone Cell Activity | 48 hours post exercise
  Bone markers (OPG, RANKL, OC) measured in serum/plasma.
Acute Bone Cell Activity | 48 hours post exercise
  Bone markers (SOST) measured in serum/plasma.
Acute Bone Cell Activity | 48 hours post exercise
  Bone markers (CTX) measured in serum/plasma.

OTHER OUTCOMES:
Inflammation | Baseline
  Interleukin 6, Interleukin 10, Interleukin 1B, TNFa measured in serum/plasma.
Inflammation | 5 minutes post exercise
  Interleukin 6, Interleukin 10, Interleukin 1B, TNFa measured in serum/plasma.
Inflammation | 1 hour post exercise
  Interleukin 6, Interleukin 10, Interleukin 1B, TNFa measured in serum/plasma.
Inflammation | 24 hour post exercise
  Interleukin 6, interleukin 10, Interleukin 1B, TNFa measured in serum/plasma.
Inflammation | 48 hour post exercise
  Interleukin 6, interleukin 10, Interleukin 1B, TNFa measured in serum/plasma.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea R Josse, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No